CLINICAL TRIAL: NCT04608318
Title: A Phase 3 Multicentre, Randomized, Prospective, Open-label Trial of Ibrutinib Monotherapy Versus Fixed-duration Venetoclax Plus Obinutuzumab Versus Fixed-duration Ibrutinib Plus Venetoclax in Patients with Previously Untreated Chronic Lymphocytic Leukaemia (CLL)
Brief Title: Ibrutinib Monotherapy Versus Fixed-duration Venetoclax Plus Obinutuzumab Versus Fixed-duration Ibrutinib Plus Venetoclax in Patients with Previously Untreated Chronic Lymphocytic Leukaemia (CLL)
Acronym: CLL17
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Stichting Hemato-Oncologie voor Volwassenen Nederland (HOVON) (Unknown); Nordic CLL Study Group (NCLLSG) (Unknown); Swiss Group for Clinical Cancer Research (SAKK) (Unknown); Cancer Trials Ireland (Network); Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) (Unknown); Grupo Español de Leucemia Linfocítica Crónica (GELLC) (Other Government); The Israeli CLL Study Group (ICLLSG) (Unknown); Janssen Pharmaceutica N.V., Belgium (Industry); AbbVie (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL17; 2022-500439-35-00 (EU CTIS Number); 2019-003854-99 (EudraCT Number)
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Chronic Lymphoid Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, B-Cell | interventions — ibrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- I (Ibrutinib) (Experimental): Ibrutinib p.o. will be administered until occurrence of unacceptable toxicity, progression of CLL or end of trial, whichever occurs first.
  Interventions: Biological: Ibrutinib
- VG (Obinutuzumab + Venetoclax) (Experimental): 12 cycles (q 28d): Obinutuzumab i.v. + Venetoclax p.o. will be administered for 6 cycles, followed by 6 additional cycles of Venetoclax alone
  Interventions: Biological: Venetoclax; Biological: Obinutuzumab
- VI (Venetoclax + Ibrutinib) (Experimental): 15 cycles (q 28d): Ibrutinib p.o. + Venetoclax p.o. will be administered for a total of 12 cycles with a prior Ibrutinib monotherapy lead-in of 3 cycles
  Interventions: Biological: Ibrutinib; Biological: Venetoclax

INTERVENTIONS:
Biological: Ibrutinib — Cycles 1 - X: 420 mg daily, d1-28 p.o.
  Other Names: Imbruvica
  Arms: I (Ibrutinib); VI (Venetoclax + Ibrutinib)
Biological: Venetoclax — Arm VG
  Cycle 1: 20 mg (2 tabl. at 10 mg), d22-28 p.o.
  Cycle 2: 50 mg (1 tabl. at 50 mg), d1-7; 100 mg (1 tabl. at 100 mg), d8-14; 200 mg (2 tabl. at 100 mg), d15-21; 400 mg (4 tabl. at 100 mg), d22-28 p.o.
  Cycles 3-12: 400 mg (4 tabl. at 100 mg), d1-28 p.o.
  Arm VI
  Cycle 4: 20 mg (2 tabl. at 10 mg), d1-7; 50 mg (1 tabl. at 50 mg), d8-14; 100 mg (1 tabl. at 100 mg), d15-21; 200 mg (2 tabl. at 100 mg), d22-28 p.o.
  Cycles 5-15: 400 mg (4 tabl. at 100 mg), d1-28 p.o.
  Other Names: ABT-199, Venclyxto
  Arms: VG (Obinutuzumab + Venetoclax); VI (Venetoclax + Ibrutinib)
Biological: Obinutuzumab — Cycle 1: (100 mg, d1 + 900 mg, d2) or 1000 mg, d1; 1000 mg, d8 + d15 i.v. Cycle 2 - 6: 1000 mg, d1 i.v.
  Other Names: GA101, Gazyvaro
  Arms: VG (Obinutuzumab + Venetoclax)

SUMMARY:
The aim of this study is to compare the efficacy of continuous ibrutinib monotherapy with fixed-duration venetoclax plus obinutuzumab and fixed-duration ibrutinib plus venetoclax by measuring progression-free survival (PFS) in patients with previously untreated CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Documented CLL requiring treatment according to iwCLL criteria.
2. Age at least 18 years.
3. Life expectancy ≥ 6 months.
4. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements.
5. Adequate bone marrow function independent of growth factor or transfusion support within 2 weeks of screening initiation as follows, unless cytopenia is due to CLL:

   1. Absolute neutrophil count ≥ 1.0 × 109/L
   2. Platelet counts ≥ 30 × 109/L; in cases of thrombocytopenia clearly due to CLL (per the discretion of the investigator), platelet count should be ≥ 10 × 109/L
   3. Total haemoglobin ≥ 8 g/dL (without transfusion support, unless anaemia is due to CLL)
6. GFR >30ml/min directly measured with 24hr urine collection, calculated according to the modified formula of Cockcroft and Gault (for men: GFR ≈ ((140 - age) x bodyweight)/ (72 x creatinine), for women x 0, 85) or an equally accurate method.

   a. For patients with creatinine values within the normal range the calculation of the clearance is not necessary. Dehydrated patients with an estimated creatinine clearance less than 30 ml/min may be eligible if a repeat estimate after adequate hydration is > 30 ml/min.
7. Adequate liver function as indicated by a total bilirubin ≤ 2 x, AST/ ALT ≤ 2.5 x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome.
8. Negative serological testing for hepatitis B (HbsAg negative and anti-HBc negative; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every month/every three months if persistently negative until 12 months after last treatment cycle), and for hepatitis C (anti-HCV-ab negative; in case of positive HCV anti-body test, negative HCV-PCR is required).
9. Eastern Cooperative Oncology Group Performance Status (ECOG) performance status 0-2.

Exclusion criteria:

1. Any prior CLL-specific therapies (except corticosteroid treatment administered due to necessary immediate intervention; within the last 10 days before start of study treatment, only dose equivalents up to 20 mg prednisolone are permitted).
2. Transformation of CLL (Richter transformation). When Richter transformation is suspected, PET-CT and/or biopsy should be performed to rule out transformation.
3. Patients with a history of PML.
4. An individual organ/ system impairment score of 4 as assessed by the CIRS definition limiting the ability to receive the study treatment or any other life-threatening illness, medical condition or organ system dysfunction that, in the investigator´s opinion, could compromise the patients' safety or interfere with the absorption or metabolism of the study drugs (e.g. inability to swallow tablets or impaired resorption in the gastrointestinal tract).
5. Malignancies other than CLL currently requiring systemic therapies, not being treated with curative intent before (unless the malignant disease is in a stable remission due to the discretion of the treating physician or showing signs of progression after curative treatment.
6. Uncontrolled or active infection.
7. Patients with known infection with human immunodeficiency virus (HIV).
8. Requirement of therapy with strong CYP3A4 and CYP3A5 inhibitors/ inducers (incl. up to 7 days prior to study treatment start).
9. Anticoagulant therapy with warfarin, phenprocoumon or other vit-amin K antagonists (alternative anticoagulation is allowed (e.g. DOACs), but patients must be properly informed about the potential risk of bleeding under treatment with ibrutinib).
10. History of stroke or intracranial hemorrhage within 6 months prior to registration for study screening.
11. Known bleeding disorders
12. Child B / C liver cirrhosis
13. Use of investigational agents which might interfere with the study drug within 28 days prior to registration for study screening.
14. Vaccination with live vaccines 28 days prior to registration for study screening.
15. Major surgery less than 30 days before start of study treatment.
16. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, known sensitivity or allergy to murine products.
17. Known hypersensitivity to any active substance or to any of the excipients of one of the drugs used in the trial.
18. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of study treatment; further pregnancy testing will be performed monthly).
19. Fertile men or women of childbearing potential unless:

    1. surgically sterile or ≥ 2 years after the onset of menopause
    2. willing to use two methods of reliable contraception including one highly effective contraceptive method (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after the end of study treatment.
20. Legal incapacity.
21. Prisoners or subjects who are institutionalized by regulatory or court order.
22. Persons who are in dependence to the sponsor or an investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 897 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed progression-free survival (PFS) | Up to 80 month
  Time from randomization to the first occurrence of progression or relapse (determined using standard iwCLL guidelines), or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Rates of undetectable minimal residual disease (uMRD) in peripheral blood (PB) and bone marrow (BM) | At final restaging (RE): 18 months after start of treatment and additional BM assessment approx. 12 months after RE
  Undetectable MRD (uMRD) is defined as <10-4 (=1 CLL-cell per 10,000 leukocytes analyzed).The uMRD rate is defined as the proportion of patients having achieved uMRD.
MRD levels in PB at different time points | Up to 80 month
  MRD is defined as the number of CLL-cells that can be detected in peripheral blood (PB) or bone marrow (BM). MRD values will be categorized into negative (<10-4) and positive (≥10-4)
Overall response rate (ORR) | At final restaging (RE): 18 months after start of treatment
  Proportion of patients having achieved a complete response (CR), a CR with incomplete recovery of the bone marrow (CRi), or a partial response (PR) as best response.
CR/CRi rate | At final restaging (RE): 18 months after start of treatment
  Proportion of patients having achieved a CR or CRi as best response (= number of patients with best response CR or CRi divided by the number of the intention-to-treat population (ITT) population)
Event-free survival | Up to 80 month
  Event-free survival (EFS) (I vs VG and I vs VI)
Time to next treatment | Up to 80 month
  Time to next treatment (TTNT)
PFS2 | Up to 80 month
  Progression free survival 2 (i.e. PFS after second-line treatment)
Incidence of safety parameters such as adverse events (AE) and adverse events of particular/special interest (AEPI/AESI) | Up to 80 month
  Type, frequency, severity and relationship to study treatment.of AEs and AEPIs/AESIs
Safety parameter TLS | Up to 80 month
  Tumour lysis syndrome (TLS) risk category after G or I lead-in (before venetoclax ramp up)

CONTACTS AND LOCATIONS:
Overall Officials: Othman Al-Sawaf, Dr. med., Principal Investigator — German CLL Study Group
Locations (181):
- Austria (5):
  - LKH-Universtitätsklinikum Graz, Graz
  - Landeskrankenhaus - Universitätskliniken Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
  - Hanusch Krankenhaus, Vienna
  - Wiener Gesundheitsverbund Klinik Ottakring, Vienna
- Belgium (3):
  - Algemeen Ziekenhuis St. Jan, Bruges
  - Universitair Ziekenhuis Leuven, Leuven
  - Algemeen Ziekenhuis Delta, Roeselare
- Denmark (8):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Regionshospitalet Holstebro, Holstebro
  - Odense Universitetshospital, Odense
  - Zealand University Hospital, Roskilde
  - Lillebaelt Vejle Sygehus, Vejle
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Germany (63):
  - Universitätsklinikum Augsburg, Augsburg
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Charite Universitaetsmedizin - Campus Benjamin Franklin, Berlin
  - Helios Klinikum Berlin Buch, Berlin
  - Charite Universitätsmedizin - Campus Virchow Klinikum, Berlin
  - Ev. Diakoniekrankenhaus, Bremen
  - Universitätsklinik Köln, Cologne
  - Gemeinschaftspraxis für Hämatologie & Onkologie, Dortmund
  - Gemeinschaftspraxis Hämatologie Onkologie, Dresden
  - Universitätsklinik Carl Gustav Carus, Dresden
  - Sana Krankenhaus Benrath, Düsseldorf
  - St. Georg Klinikum Eisenach, Eisenach
  - ISP Erlangen Onkologische Schwerpunktpraxis, Erlangen
  - Universitätsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Onkologische Schwerpunktpraxis, Esslingen am Neckar
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Uniklinikum Gießen und Marburg, Giessen
  - MVZ Onkologische Kooperation Harz, Goslar
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - OncoResearch Lerchenfeld, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Onkologisches Ambulanzzentrum - MediProjekt, Hanover
  - Onkologische Schwerpunktpraxis Heidelberg, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Marien Hospital Herne, Herne
  - Universitätskliniken des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Praxis für Haematologie und Onkologie, Koblenz
  - MVZ Hämatologie Onkologie Koblenz, Koblenz
  - H.O.T Onkologie Praxis Landshut, Landshut
  - Universitätsklinikum Leipzig, Leipzig
  - Onkopraxis Probstheida, Leipzig
  - Klinikum Lippe Lemgo, Lemgo
  - St Vincenz Krankenhaus, Limburg
  - Lübecker Onkologische Schwerpunktpraxis, Lübeck
  - Gemeinschaftspraxis Haematologie und Onkologie, Magdeburg
  - Universitätsklinikum Magdeburg, Magdeburg
  - Mannheimer Onkologie Praxis, Mannheim
  - Praxis für Innere Medizin - Hämatologie und Onkologie, Marburg
  - Kliniken Maria Hilf, Mönchengladbach
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - München Klinik Schwabing, München
  - Klinikum der Universitaet München - Grosshadern Campus, München
  - Klinikum rechts der Isar - Technische Universitaet Muenchen, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Klinikum Oldenburg, Oldenburg
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Ravensburg
  - Barmherzigen Brüder Krankenhaus, Regensburg
  - Schwerpunktpraxis für Hämatologie & Onkologie - OncoPro GbR, Regensburg
  - Universitätsklinik Rostock, Rostock
  - OnkoSaar Praxis für Hämatologie und Onkologie, Saarbrücken
  - Zentrum für abulante Hämatologie und Onkologie, Siegburg
  - Marienhospital Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - MVZ Weiden GmbH, Weiden
  - Hämatologisch Onkologische Schwerpunktpraxis, Würzburg
- Ireland (8):
  - Cork University Hospital, Cork
  - St Vincents University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford
- Israel (10):
  - Soroka University Medical Center, Beersheba
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Bnai-Zion Medical Center, Haifa
  - Hadassah Medical Center Ein Kerem University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Ospedale dell'Angelo, Mestre
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale S. Maria della Misericordia, Perugia
  - Umberto I - Policlinico di Roma - Sapienza Università, Roma
  - Gmelli University Hospital, Roma
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino, Torino
- Netherlands (22):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Nordwest Ziekenhuisgroep, Locatie Alkmaar, Alkmaar
  - OLVG Amsterdam, Amsterdam
  - Amsterdam Universitair Medische Centra, Amsterdam
  - Rijnstate, Locatie Arnhem, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Ziekenhuis, Delft
  - Slingeland ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Martini Ziekenhuis, Groningen
  - Ziekenhuis St Jansdal, Harderwijk
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, Leiderdorp
  - St. Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
  - Franciscus Vlietland, Schiedam
  - Ziekenhuis Rivierenland Tiel, Tiel
  - Diakonessenhuis, Utrecht
  - VieCuri Medish Centrum, Venlo
  - Isala Zwolle, Zwolle
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - St. Olavs Hospital Trondheim University Hospital, Trondheim
- Spain (15):
  - Hospital Germans Trias i Pujol, Badalona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Costa del Sol, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Marques de Valdecilla, Santander
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clinico Universitario Valencia, Valencia
  - Residencia Sanitaria La Fe - Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Sweden (12):
  - Soedra Aelvsborgs Sjukhus, Borås
  - Falu Lasarett, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Hallands Sjukhus Halmstad, Halmstad
  - Universitetssjukhuset Linköping, Linköping
  - Sunderby Hospital, Luleå
  - Skåne University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital Solna, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Hallands Sjukhus, Varberg
- Switzerland (18):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Oberwallis, Brig
  - Kantonsspital Graubünden, Chur
  - HFR Fribourg Hôpital cantonal, Fribourg
  - Hôpitaux Universitaires Genève, Geneva
  - Kantonsspital Baselland, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Spital Thurgau AG - Kantonsspital Münsterlingen, Münsterlingen
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital Thun, Thun
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - Universitätsspital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Sawaf O, Stumpf J, Zhang C, Simon F, Bosch F, Feyzi E, Ghia P, Gregor M, Kater AP, Lindstrom V, Mattsson M, Niemann CU, Staber PB, Tadmor T, Thornton P, Wendtner CM, Janssens A, Noesslinger T, Bohn JP, da Cunha-Bang C, Poulsen CB, Ranti J, Illmer T, Schoettker B, Bottcher S, Gaska T, Vandenberghe E, Clifford R, Benjamini O, Frustaci AM, Scarfo L, Sportoletti P, Schreurs J, Levin MD, van der Straaten H, van der Klift M, Tran H, de la Serna J, Loscertales J, Lindblad O, Bergendahl Sandstedt A, Goede J, Baumann M, Fink AM, Fischer K, Ritgen M, Kreuzer KA, Schneider C, Tausch E, Stilgenbauer S, Robrecht S, Eichhorst B, Hallek M; CLL17 Trial Investigators. Fixed-Duration versus Continuous Treatment for Chronic Lymphocytic Leukemia. N Engl J Med. 2025 Dec 6. doi: 10.1056/NEJMoa2515458. Online ahead of print. PMID 41358601
- See also: Click here for more information about this study: CLL17 (German CLL Study Group) — https://www.dcllsg.com/cll17/